CLINICAL TRIAL: NCT03465332
Title: Use of Diagnostic Measures (Including Blood Eosinophil Counts) and Their Impact on Lung Specialists' Treatment Decisions in Patients With COPD in Germany
Brief Title: Use of Diagnostic Measures in Chronic Obstructive Pulmonary Disease (COPD) in Routine Practice and Their Impact on Treatment Decisions
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Institut Dr. Schauerte (IDS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 207733
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: blood eosinophil count; COPD; diagnostic test; doctor's questionnaire; Lung specialist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung specialist: Approximately 30 lung specialists in Germany with a sufficient number of COPD subjects under supervision will be enrolled in the study to document physician's attitudes on COPD diagnosis and therapy, and to document data on about 250 subjects with COPD.
  Interventions: Other: Doctor's questionnaire
- Subjects with COPD: Data from approximately 250 subjects with COPD under supervision of lung specialists enrolled in the study will be analyzed.
  Interventions: Other: Subject file

INTERVENTIONS:
Other: Doctor's questionnaire — The survey of physicians will be performed using doctor's questionnaire, which will be developed by lung specialists who are not participating in the survey.
  Groups: Lung specialist
Other: Subject file — All subject-based data will be obtained by retrospective evaluation of subject files available at the treating lung specialist.
  Groups: Subjects with COPD

SUMMARY:
This study will evaluate the diagnostic measures (including blood eosinophil counts) commonly used by lung specialist's in routine clinical care of subjects with COPD in Germany and how these diagnostic tests influence the physician's treatment decisions. The study will be conducted in three parts. In the first part, lung specialist's, who will not participate in the survey, will develop doctor's questionnaire. The second part is an interventional cross-sectional study, wherein approximately 30 lung specialists will be enrolled and data on their perspective on diagnosis and treatment of COPD subjects will be collected via the revised doctor's questionnaire. The third part is a retrospective non-interventional study where each doctor will collect retrospective data from selected subjects with COPD from the time of informed consent up to 12 months before. The retrospective data will be collected from subject files of approximately 250 subjects with COPD.

ELIGIBILITY:
Inclusion Criteria:

For participating centers (Sample 1: 30 lung specialists from Germany)

* More than 10 years of experience in respiratory medicine
* At least 500 subjects under supervision in hospital- or office-based setting: a) Focus on obstructive lung diseases. b) Board certification. c) Informed consent to participate in this study and to share files of consenting subjects.

For subjects (Sample 2: 250 COPD subjects from these 30 doctors from sample 1)

* Written informed consent to use his/her data.
* Age >=40 years
* Pack years >10, current or former smoking
* Duration of COPD: >=1 year since COPD diagnosis record in subject files (also confirmed by spirometry)
* No concurrent asthma diagnosis
* At least one year of documented disease history at participating study doctors and have to be under the care of the before mentioned physician during this time because of COPD.

Exclusion Criteria:

* Subjects who are pregnant and breastfeeding (in the last 12 months)
* Subjects currently participating in any interventional study
* Subjects with severe comorbidities which would have influence on the COPD therapy

Min Age: 35 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Approximately 30 lung specialists (up to 50) in Germany with sufficient number of COPD subjects under supervision in a hospital or office based setting will be enrolled in the study. Data from the survey of lung specialists and retrospective medical data of 250 subjects with COPD under supervision of the 30 lung specialists (up to 50) enrolled in the study will be included in the analysis.
Sampling Method: Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Number of physicians with usage of diagnostic tests in routine clinical practice | Up to 12 months
  The data on diagnostic test including blood eosinophil count commonly used by lung specialists in routine clinical practice will be obtained from doctor's questionnaire.
Number of physician reported rationale for choice of diagnostic test | Up to 12 months
  The reasons for choice of diagnostic test will be determined from doctor's questionnaires and from medical chart review.

SECONDARY OUTCOMES:
Number of physician reported reasons for blood eosinophil test selection | Up to 12 months
  The reasons blood eosinophil test selection will be analyzed using data from doctor's questionnaires.
Number of physician reported reasons for drug selection | Up to 12 months
  The selection of drugs by lung specialists for subjects with COPD will be analyzed using information obtained from medical chart review.
Number of subjects with use of other diagnostic measures | Up to 12 months
  Number of subjects with use of other diagnostic measures such as spirometry, X-ray, thoracic computer tomography and specific blood tests will be analyzed using data from subject files.
Number of subjects with use of patient reported outcome (PRO) assessment | Up to 12 months
  Number of subjects with use of questionnaires like COPD assessment test (CAT) and dyspnea assessment will be analyzed using data from subject files.
Number of subjects with a history of respiratory medication | Up to 12 months
  Number of subjects with a history of respiratory medication will be analyzed using data from subject files.
Number of subjects receiving current medication | Up to 12 months
  Number of subjects receiving current medication will be analyzed using data from subject files.
Number of subjects receiving COPD maintenance treatment | Up to 12 months
  Number of subjects receiving COPD maintenance treatment will be analyzed using data from subject files.
Number of subjects receiving immunosuppressive treatment | Up to 12 months
  Number of subjects receiving immunosuppressive treatment will be analyzed using data from subject files.
Number of subjects receiving allergic treatment | Up to 12 months
  Number of subjects receiving allergic treatment will be analyzed using data from subject files.
Number of subjects receiving oral corticosteroids (OCS) for exacerbations | Up to 12 months
  Number of subjects with maintenance and rescue use of OCS for exacerbations will be analyzed using data from subject files.
Number of subjects with use of antibiotics | Up to 12 months
  Number of subjects with use of antibiotics will be analyzed using data from subject files.
Number of subjects receiving any COPD medication | Up to 12 months
  Number of subjects receiving any COPD medication will be analyzed using data from subject files.
Number of subjects with history of exacerbations | Up to 12 months
  Number of subjects with history of exacerbations will be analyzed using data from subject files.
Number of subjects with hospitalization for COPD | Up to 12 months
  Number of subjects with hospitalization for COPD will be analyzed using data from subject files.
Number of subjects with emergency room visits related to COPD | Up to 12 months
  Number of subjects with emergency room visits related to COPD will be analyzed using data from subject files.
Number of subjects with concomitant diseases | Up to 12 months
  Number of subjects with concomitant diseases will be analyzed using data from subject files.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (23):
- Germany (23):
  - GSK Investigational Site, Bruchsal, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Garmisch-Partenirchen, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Beelitz, Brandenburg
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Fürstenwalde, Brandenburg
  - GSK Investigational Site, Kyritz, Brandenburg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Gütersloh, North Rhine-Westphalia
  - GSK Investigational Site, Menden, North Rhine-Westphalia
  - GSK Investigational Site, Warendorf, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halberstadt, Saxony-Anhalt
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Hettstedt, Saxony-Anhalt
  - GSK Investigational Site, Wittenberg, Saxony-Anhalt
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: No